CLINICAL TRIAL: NCT06341400
Title: Perioperative Efficacy of RC48 Combined with Toripalimab in Treatment of Cisplatin Ineligible MIBC
Brief Title: RC48 Combined with Toripalimab As Neoadjuvant Therapy for Cisplatin Ineligible MIBC Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Abai Xu, Chief, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-030-01
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-09

CONDITIONS: Bladder Cancer; Muscle-Invasive Bladder Carcinoma
Keywords: Neoadjuvant Therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Each subject will receive RC48-ADC 2.0mg/kg and toripalimab 3.0mg/kg intravenously every 2 weeks for a total of 4 cycles. RC48-ADC 2.0mg/kg and toripalimab 3.0mg/kg were intravenously infused every 2 weeks for 8 cycles.
  Interventions: Drug: DisitamabVedotinForIicction Toripalimab

INTERVENTIONS:
Drug: DisitamabVedotinForIicction Toripalimab — Each subject will receive RC48-ADC 2.0mg/kg and toripalimab 3.0mg/kg intravenously every 2 weeks for a total of 4 cycles. RC48-ADC 2.0mg/kg and toripalimab 3.0mg/kg were intravenously infused every 2 weeks for 8 cycles.
  Other Names: radical cystectomy

SUMMARY:
A single-arm, prospective, exploratory clinical trial to explore the pathological complete response (pCR) rate of immune checkpoint inhibitors combined with antibody conjugate drugs as the perioperative treatment of platinum-intolerant bladder cancer patients. Fifty-five patients with clinically or pathologically confirmed muscle-invasive bladder urothelial carcinoma (MIBC) who were ineligible for cisplatin-based chemotherapy or refused cisplatin-based chemotherapy were enrolled. Each subject will receive RC48-ADC and toripalimab intravenously every 2 weeks for a total of 4 cycles before surgery, 8 cycles after surgery. The efficacy was evaluated and followed up after 4 cycles of neoadjuvant therapy, 3 months postoperative, and every 3-6 months thereafter. The primary endpoint of this study was pathological complete response rate (pCR). The secondary endpoints were to explore the safety, disease-free survival (DFS), overall survival (OS), objective response rate (ORR) and disease control rate (DCR) of RC48 combined with toripalimab neoadjuvant therapy followed by radical cystectomy.

DETAILED DESCRIPTION:
This study was a single-arm, prospective, exploratory clinical trial to explore the pathological complete response (pCR) rate of immune checkpoint inhibitors combined with antibody conjugate drugs as the perioperative treatment of platinum-intolerant bladder cancer patients. Fifty-five patients with clinically or pathologically confirmed muscle-invasive bladder urothelial carcinoma (MIBC) who were ineligible for cisplatin-based chemotherapy or refused cisplatin-based chemotherapy were enrolled. Each subject will receive RC48-ADC 2.0mg/kg and toripalimab 3.0mg/kg intravenously every 2 weeks for a total of 4 cycles before surgery. RC48-ADC 2.0mg/kg and toripalimab 3.0mg/kg were intravenously infused every 2 weeks for 8 cycles after surgery. The efficacy was evaluated and followed up after 4 cycles of neoadjuvant therapy, 3 months postoperative, and every 3-6 months thereafter. The primary endpoint of this study was pathological complete response rate (pCR). The secondary endpoints were to explore the safety, disease-free survival (DFS), overall survival (OS), objective response rate (ORR) and disease control rate (DCR) of RC48 combined with toripalimab neoadjuvant therapy followed by radical cystectomy. In the process of research, plasma and tumor tissues need to be obtained for proteomics and genomics analysis to explore the relationship between potential predictive biomarkers and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to provide written informed consent.
2. Male or female, aged ≥18 years old.
3. Patients must be ineligible for cisplatin-based chemotherapy or refuse cisplatin-based chemotherapy because of any of the following:

   Creatinine clearance (CrCl) <60 mL/min, ECOG performance status (PS) 0-1 Creatinine clearance (CrCl) ≥ 60 mL/min, ECOG PS 2 (if the patient is eligible for RC) Hearing impairment ≥ CTCAE level 2 According to CTCAE criteria, neuropathy was ≥ grade 2 The patient declined cisplatin-based chemotherapy
4. Patients must be medically suitable for TURBT and RC.
5. Pathological examination and immunohistochemical Her-2 (≥1+)
6. measurable lesions according to RECIST 1.1.
7. Adequate organ function, as demonstrated by the following laboratory results within 7 days before study treatment:

   The heart ejection fraction was ≥50%. Hemoglobin ≥9 g/dL; Absolute neutrophil count ≥ 1.5×109 /L and platelet ≥ 100×109 /L; Total bilirubin ≤ 1.5× ULN; AST and ALT ≤ 2.5×ULN and ≤ 5×ULN.
8. All female subjects will be considered to be of reproductive potential unless they are postmenopausal or have been surgically sterilized. Female subjects of childbearing potential had to consent to the use of highly effective contraception. Male subjects of childbearing potential and their female partners had to consent to the use of highly effective contraception.
9. Be willing to comply with the study access schedule and the prohibitions and restrictions set forth in this Agreement.

Exclusion Criteria:

1. known hypersensitivity to components of recombinant humanized anti-HER2 monoclonal antibody-MMAE conjugate or allergic reaction to toripalimab.
2. toxicity from previous antineoplastic therapy did not revert to CTCAE grade 0-1 (except grade 2 alopecia).
3. pleural or abdominal effusion with clinical symptoms requiring ongoing treatment.
4. history of major surgery within 4 weeks of planned initiation of trial treatment.
5. received live virus vaccine within 4 weeks after planned initiation of trial treatment.
6. currently known active HIV or tuberculosis infection.
7. diagnosed as HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive.
8. there is history or current evidence of any condition, treatment, or laboratory abnormality that the treatment investigator believes may confound the trial results, interfere with the participant's participation throughout the trial, or be inconsistent with the participant's participation.
9. history of other malignancies within the past 5 years.
10. known central nervous system metastases
11. uncontrolled hypertension, diabetes, interstitial lung disease, or chronic obstructive pulmonary disease.
12. receiving systemic therapy (e.g., immunomodulatory agents, corticosteroids, or immunosuppressive agents) for autoimmune disease within 2 years before study treatment.
13. NYHA class III heart failure.
14. pregnancy or lactation.
15. were assessed by the investigator as unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
PcR | 2months
  The resected primary tumor specimen and all sampled regional lymph nodes (ypT0N0) had no viable tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Abai Xu, doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China